CLINICAL TRIAL: NCT02452034
Title: A Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous (IV) and Powder for Oral Suspension Formulations of Posaconazole (POS) in Immunocompromised Pediatric Subjects With Neutropenia
Brief Title: Safety and Pharmacokinetics of Intravenous and Oral Posaconazole in Immunocompromised Children (MK-5592-097)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5592-097; 2014-002807-10 (EudraCT Number); MK-5592-097 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Neutropenia
MeSH Terms: conditions — Neutropenia | interventions — posaconazole; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 3.5 mg/kg POS (2<7 years old) (Experimental): Children 2 to less than 7 years of age will receive POS at 3.5 mg/kg by intravenous (IV) solution twice on Day 1, then once daily on Days 2-10. This will be followed by treatment with 3.5 mg/kg POS once daily by powder for oral suspension (PFS) for a minimum of 10 days; or, if they are unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
  Interventions: Drug: Posaconazole IV solution; Drug: Posaconazole powder for oral suspension
- 4.5 mg/kg POS (2<7 years old) (Experimental): Children 2 to less than 7 years of age will receive POS at 4.5 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This will be followed by treatment with 4.5 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they are unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
  Interventions: Drug: Posaconazole IV solution; Drug: Posaconazole powder for oral suspension
- 3.5 mg/kg POS (7-17 years old) (Experimental): Children 7 to 17 years of age will receive POS at 3.5 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This will be followed by treatment with 3.5 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they are unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
  Interventions: Drug: Posaconazole IV solution; Drug: Posaconazole powder for oral suspension
- 4.5 mg/kg POS (7-17 years old) (Experimental): Children 7 to 17 years of age will receive POS at 4.5 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This will be followed by treatment with 4.5 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they are unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
  Interventions: Drug: Posaconazole IV solution; Drug: Posaconazole powder for oral suspension
- 6 mg/kg POS (2<7 years old) (Experimental): Children 2 to less than 7 years of age will receive POS at 6 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This will be followed by treatment with 6 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they are unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
  Interventions: Drug: Posaconazole IV solution; Drug: Posaconazole powder for oral suspension
- 6 mg/kg POS (7-17 years old) (Experimental): Children 7 to 17 years of age will receive POS at 6 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This will be followed by treatment with 6 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they are unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
  Interventions: Drug: Posaconazole IV solution; Drug: Posaconazole powder for oral suspension

INTERVENTIONS:
Drug: Posaconazole IV solution — Posaconazole by IV solution twice on Day 1, then once daily on Days 2-10.
  Other Names: Noxafil
Drug: Posaconazole powder for oral suspension — Posaconazole once daily by PFS for a minimum of 10 days
  Other Names: Noxafil

SUMMARY:
This study aims to evaluate the pharmacokinetics of posaconazole (POS) administered intravenously (IV) or orally to immunocompromised pediatric participants.

ELIGIBILITY:
Inclusion Criteria:

* Have documented or anticipated neutropenia expected to last for at least 7 days, following treatment in at least one of the following clinical situations: acute leukemia, myelodysplasia, severe aplastic anemia, recipients of Autologous Hematopoietic Stem Cell Transplant (HSCT), high risk neuroblastoma, advanced stage non-Hodgkin's lymphoma, hemophagocytic lymphohistiocytosis
* Have a central line in place prior to IV study therapy
* Participants of reproductive potential agree to remain abstinent, or use a medically accepted method of birth control

Exclusion Criteria:

* Has a proven or probable invasive fungal infection
* Has received any formulation of POS within prior 10 days
* Is receiving any prohibited drugs
* Has laboratory results that are outside of normal limits at screening, as follows: a) Moderate or severe liver dysfunction, as defined as: Aspartate Aminotransferase (AST) > 5 times the upper limit of normal (ULN), OR Alanine Aminotransferase (ALT) > 5 times the ULN, OR Serum total bilirubin >2.5 times the ULN, OR AST or ALT > 3 times ULN with total bilirubin > 2 times ULN; b) Calculated creatinine clearance <30 mL/min.
* Has QTc (QT interval corrected for rate) prolongation defined as: a) Symptomatic QTc prolongation >450 msec (males) or >470 msec (females) OR b) Any QTc prolongation of >500 msec
* Is pregnant, intends to become pregnant during study, or is breastfeeding
* Has a history of anaphylaxis attributed to the azole class of antifungal agents
* Is not expected to receive a minimum of 10 days of POS IV solution
* Has participated in any Phase 1 Investigational New Drug (IND) study within prior 30 days or expects to do so within the following 60 days
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Groll AH, Abdel-Azim H, Lehrnbecher T, Steinbach WJ, Paschke A, Mangin E, Winchell GA, Waskin H, Bruno CJ. Pharmacokinetics and safety of posaconazole intravenous solution and powder for oral suspension in children with neutropenia: an open-label, sequential dose-escalation trial. Int J Antimicrob Agents. 2020 Sep;56(3):106084. doi: 10.1016/j.ijantimicag.2020.106084. Epub 2020 Jul 17. PMID 32682946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Immunocompromised participants aged 2 to 17 years old, with neutropenia expected to last for at least 7 days following start of study treatment, were enrolled in this study.
Groups:
- 3.5 mg/kg POS (2<7 Years Old): Children 2 to less than 7 years of age received posaconazole (POS) at 3.5 mg/kg by intravenous (IV) solution twice on Day 1, then once daily on Days 2-10. This was followed by treatment with 3.5 mg/kg POS once daily by powder for oral suspension (PFS) for a minimum of 10 days; or, if they were unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
- 3.5 mg/kg POS (7-17 Years Old): Children 7 to 17 years of age received POS at 3.5 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This was followed by treatment with 3.5 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they were unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
- 4.5 mg/kg POS (2<7 Years Old): Children 2 to less than 7 years of age received POS at 4.5 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This was followed by treatment with 4.5 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they were unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
- 4.5 mg/kg POS (7-17 Years Old): Children 7 to 17 years of age received POS at 4.5 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This was followed by treatment with 4.5 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they were unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
- 6 mg/kg POS (2<7 Years Old): Children 2 to less than 7 years of age received POS at 6 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This was followed by treatment with 6 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they were unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
- 6 mg/kg POS (7-17 Years Old): Children 7 to 17 years of age received POS at 6 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This was followed by treatment with 6 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they were unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
Period: Overall Study
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old)
Started | 16 | 21 | 15 | 17 | 20 | 29
Treated | 14 | 21 | 15 | 16 | 20 | 29
Completed | 14 | 20 | 14 | 16 | 19 | 26
Not Completed | 2 | 1 | 1 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Screen Failure | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawn by Parent/Guardian | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old) | Total
Number analyzed (Participants) | 16 | 21 | 15 | 17 | 20 | 29 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.9 (1.5) | 13.9 (2.1) | 4.1 (1.4) | 12.5 (2.7) | 3.9 (1.6) | 12.0 (3.5) | 8.9 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 8 | 8 | 10 | 10 | 50
  Male | 13 | 10 | 7 | 9 | 10 | 19 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 4 | 1 | 2 | 12
  Not Hispanic or Latino | 15 | 19 | 12 | 12 | 18 | 27 | 103
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 1 | 2 | 2 | 1 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 2 | 3
  White | 12 | 18 | 12 | 13 | 18 | 26 | 99
  More than one race | 0 | 2 | 0 | 2 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to 24 Hours Post-dose for POS
Description: Blood was collected from pre-dose up to 24 hours post-dose in order to determine the plasma AUC from time 0-24 hours post-dose (AUC0-24hr) of posaconazole. A non compartmental analysis of posaconazole plasma concentrations was performed. Results are reported for each treatment arm according to the formulation that participants received (IV or PFS). Participants receiving both formulations were counted once for each formulation.
Time Frame: Any day from Day 7 to Day 10 of therapy for each formulation (up to 28 days) at pre-dose, within 15 minutes after end of infusion (up to 2 hours), and 4, 6, 8, 12, 24 hours post-infusion
Population: All treated participants who received at least 7 days of POS dosing (IV and PFS), completed the full POS PK sampling, and met pre-specifiied acceptability criteria.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old)
Number analyzed (Participants) | 11 | 19 | 14 | 15 | 17 | 24
hr*ng/mL
  IV | 17800 (55.0) | 27300 (49.7) | 25600 (30.0) | 29800 (42.9) | 31100 (48.9) | 44200 (41.5)
  PFS: number analyzed (Participants) | 5 | 10 | 8 | 8 | 7 | 12
  PFS | 12200 (36.0) | 20700 (33.8) | 21600 (64.5) | 28700 (33.7) | 23000 (47.3) | 25000 (184.3)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for POS
Description: Blood was collected from pre-dose up to 24 hours post-dose in order to determine the plasma Cmax of posaconazole. A non-compartmental analysis of posaconazole plasma concentrations was performed. Results are reported for each treatment arm according to the formulation that participants received (IV or PFS). Participants receiving both formulations were counted once for each formulation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old)
Number analyzed (Participants) | 11 | 19 | 14 | 15 | 17 | 24
ng/mL
  IV | 1590 (43.1) | 2450 (72.7) | 2320 (39.8) | 2310 (40.3) | 3060 (54.1) | 3340 (39.4)
  PFS: number analyzed (Participants) | 5 | 10 | 8 | 8 | 7 | 12
  PFS | 884 (44.4) | 1340 (30.8) | 1550 (40.8) | 1670 (28.5) | 1510 (43.4) | 1370 (178.5)

3. Primary Outcome: Minimum Plasma Concentration (Cmin) for POS
Description: Blood was collected from pre-dose up to 24 hours post-dose in order to determine the plasma Cmin of posaconazole. A non-compartmental analysis of posaconazole plasma concentrations was performed. Results are reported for each treatment arm according to the formulation that participants received (IV or PFS). Participants receiving both formulations were counted once for each formulation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old)
Number analyzed (Participants) | 11 | 19 | 14 | 15 | 17 | 24
ng/mL
  IV | 400 (81.3) | 670 (65.1) | 501 (56.8) | 737 (66.0) | 626 (104.8) | 1160 (60.4)
  PFS: number analyzed (Participants) | 5 | 10 | 8 | 8 | 7 | 12
  PFS | 254 (45.6) | 579 (44.9) | 476 (164.6) | 790 (48.2) | 542 (68.8) | 713 (300.6)

4. Primary Outcome: Average Steady-state Plasma Concentration (Cavg) for POS
Description: Blood was collected from pre-dose up to 24 hours post-dose in order to determine the plasma Cavg of posaconazole. A non-compartmental analysis of posaconazole plasma concentrations was performed. Results are reported for each treatment arm according to the formulation that participants received (IV or PFS). Participants receiving both formulations were counted once for each formulation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old)
Number analyzed (Participants) | 11 | 19 | 14 | 15 | 17 | 24
ng/mL
  IV | 743 (55.0) | 1140 (49.7) | 1070 (30.0) | 1240 (42.9) | 1300 (48.9) | 1840 (41.5)
  PFS: number analyzed (Participants) | 5 | 10 | 8 | 8 | 7 | 12
  PFS | 510 (36.0) | 861 (33.8) | 901 (64.5) | 1200 (33.7) | 960 (47.3) | 1040 (184.3)

5. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) for POS
Description: Blood was collected from pre-dose up to 24 hours post-dose in order to determine the plasma Tmax of posaconazole. A non-compartmental analysis of posaconazole plasma concentrations was performed. Results are reported for each treatment arm according to the formulation that participants received (IV or PFS). Participants receiving both formulations were counted once for each formulation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old)
Number analyzed (Participants) | 11 | 19 | 14 | 15 | 17 | 24
Hours
  IV | 1.78 [1.67 to 5.53] | 1.77 [0.00 to 3.50] | 1.78 [1.42 to 5.90] | 1.75 [1.52 to 1.80] | 1.75 [1.57 to 1.83] | 1.77 [1.33 to 6.00]
  PFS: number analyzed (Participants) | 5 | 10 | 8 | 8 | 7 | 12
  PFS | 3.83 [1.92 to 4.25] | 2.20 [1.92 to 6.03] | 3.82 [1.88 to 5.92] | 6.14 [1.98 to 7.98] | 4.00 [2.17 to 7.92] | 2.78 [0.00 to 4.00]

6. Primary Outcome: Total Body Clearance (CL) for POS Administered by IV
Description: Blood was collected from pre-dose up to 24 hours post-dose in order to determine the plasma CL of posaconazole administered by IV. A non-compartmental analysis of posaconazole plasma concentrations was performed. Results are reported for participants that received IV treatment.
Time Frame: Any day from Day 7 to Day 10 of therapy (up to 28 days) at pre-dose, within 15 minutes after end of infusion (up to 2 hours), and 4, 6, 8, 12, 24 hours post-infusion
Population: All treated participants who received at least 7 days of POS IV solution therapy, completed the full POS PK sampling while on POS IV solution, and met pre-specified acceptability criteria.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old)
Number analyzed (Participants) | 11 | 19 | 14 | 15 | 17 | 24
L/hr | 3.39 (52.8) | 6.64 (38.6) | 2.97 (36.2) | 6.69 (37.3) | 3.27 (49.3) | 4.76 (55.7)

7. Primary Outcome: Apparent Total Body Clearance (CL/F) for POS Administered by PFS
Description: Blood was collected from pre-dose up to 24 hours post-dose in order to determine the plasma CL/F of posaconazole administered by PFS. A non-compartmental analysis of posaconazole plasma concentrations was performed. Results are reported for participants that received PFS treatment.
Time Frame: as for outcome 6
Population: All treated participants who received at least 7 days of POS PFS therapy, completed the full POS PK sampling while on POS PFS, and met pre-specified acceptability criteria.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old)
Number analyzed (Participants) | 5 | 10 | 8 | 8 | 7 | 12
L/hr | 4.97 (29.1) | 7.67 (39.9) | 3.49 (59.1) | 7.84 (49.4) | 4.60 (35.2) | 8.39 (190.3)

8. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol - specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: 14 days after end of treatment (Up to 42 days)
Population: All participants who received at least one dose of study drug. Data were analysed as pre-specified in the study protocol, based on age group and dosage, and did not distinguish oral from IV formulation.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old)
Number analyzed (Participants) | 14 | 21 | 15 | 16 | 20 | 29
Participants | 13 | 21 | 15 | 16 | 19 | 29

9. Secondary Outcome: Number of Participants Who Discontinued Treatment of Study Drug Due to an Adverse Event (AE)
Description: as for outcome 8
Time Frame: Up to 28 days
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6 mg/kg POS (2<7 Years Old) | 6 mg/kg POS (7-17 Years Old)
Number analyzed (Participants) | 14 | 21 | 15 | 16 | 20 | 29
Participants | 3 | 3 | 0 | 2 | 4 | 6

ADVERSE EVENTS:
Time Frame: AEs and SAEs: 14 days after end of treatment (up to day 42); All-Cause Mortality: Up to day 110.
Description: All participants who received at least one dose of study drug. Participants were followed for survival up to 110 days, and deaths that occurred outside of the AE collection time frame were recorded in the Participant Flow. Data were analysed as pre-specified in the study protocol, based on age group and dosage, and did not distinguish oral from IV formulation.
Groups:
- 6.0 mg/kg POS (2<7 Years Old): Children 2 to less than 7 years of age received POS at 6 mg/kg by intravenous (IV) solution twice on Day 1, then once daily on Days 2-10. This was followed by treatment with 6 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they were unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
- 6.0 mg/kg POS (7-17 Years Old): Children 7 to 17 years of age received POS at 6 mg/kg by IV solution twice on Day 1, then once daily on Days 2-10. This was followed by treatment with 6 mg/kg POS once daily by PFS for a minimum of 10 days; or, if they were unwilling or unable to tolerate POS PFS, continued treatment with POS IV.
Arm/Group | 3.5 mg/kg POS (2<7 Years Old) | 3.5 mg/kg POS (7-17 Years Old) | 4.5 mg/kg POS (2<7 Years Old) | 4.5 mg/kg POS (7-17 Years Old) | 6.0 mg/kg POS (2<7 Years Old) | 6.0 mg/kg POS (7-17 Years Old)
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/21 | 0/15 | 0/16 | 1/20 | 2/29
Serious Adverse Events (participants affected / at risk) | 3/14 | 8/21 | 4/15 | 5/16 | 3/20 | 8/29
Other Adverse Events (participants affected / at risk) | 13/14 | 20/21 | 15/15 | 16/16 | 19/20 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.5 mg/kg POS (2<7 Years Old) (N=14) | 3.5 mg/kg POS (7-17 Years Old) (N=21) | 4.5 mg/kg POS (2<7 Years Old) (N=15) | 4.5 mg/kg POS (7-17 Years Old) (N=16) | 6.0 mg/kg POS (2<7 Years Old) (N=20) | 6.0 mg/kg POS (7-17 Years Old) (N=29)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Engraftment syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic mycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venoocclusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.5 mg/kg POS (2<7 Years Old) (N=14) | 3.5 mg/kg POS (7-17 Years Old) (N=21) | 4.5 mg/kg POS (2<7 Years Old) (N=15) | 4.5 mg/kg POS (7-17 Years Old) (N=16) | 6.0 mg/kg POS (2<7 Years Old) (N=20) | 6.0 mg/kg POS (7-17 Years Old) (N=29)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (4) | 1 (1) | 1 (2) | 3 (4) | 2 (2) | 2 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 7 (7) | 7 (8)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (3) | 2 (4)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 6 (8) | 2 (2) | 5 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 5 (5) | 4 (4) | 5 (6) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (5) | 1 (1) | 3 (5) | 2 (2) | 7 (9)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oral mucosal exfoliation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scalloped tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 6 (6)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (6) | 6 (9) | 2 (3) | 6 (8) | 6 (8) | 6 (13)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mucosal inflammation (General disorders) | 3 (3) | 9 (10) | 5 (5) | 4 (4) | 5 (5) | 6 (6)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (13) | 9 (11) | 6 (9) | 10 (13) | 8 (8) | 8 (12)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Engraftment syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Graft versus host disease (Immune system disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Immunodeficiency (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immunodeficiency common variable (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum sickness (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BK virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Human bocavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Buttock injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (6)
BK polyomavirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood culture positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug level increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid balance positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Pulmonary arterial pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Viral test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 3 (3) | 1 (1) | 3 (3) | 4 (4)
Fluid intake reduced (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 7 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Magnesium deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (2) | 3 (5) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0) | 5 (6) | 1 (1) | 5 (7)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intention tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Opisthotonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 1 (1) | 5 (8) | 1 (1) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar exudate (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 4 (5) | 7 (7)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4) | 3 (4) | 2 (2) | 4 (6) | 3 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 2 (2) | 2 (2) | 1 (1) | 6 (6) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venoocclusive disease (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT02452034/Prot_SAP_000.pdf